Title: Addressing Social Determinants of Health to Reduce Physician Burnout

NCT04070456 Date: 11/5/2019 You are invited to participate in a research study (IRB #00059798). Physician and care team well-being are important to a health organization. We are pleased to collaborate with the American Medical Association (AMA) to conduct this survey and advance strategies that restore joy, purpose, and meaning to clinicians and care teams, which improving healthcare delivery and quality outcomes for our patients. Your participation in this research will involve completing this survey three times (baseline, 6 months, and 12 months).

The purpose of this study is to evaluate if addressing patients' unmet social needs improves clinician burnout. You are invited to be in this study because you are a clinician at one of the participating clinic sites. Your participation in this study is voluntary. Up to 80 clinicians will take part in this study. You do not have to participate in this study if you do not want to, and we will keep all of your responses private and confidential. There is no specific benefit to you for participating in this study. There are no costs to you associated with participating in the study and any study costs, related directly to the study, will be paid for by the study. You will receive no payment or other compensation for taking part in this study.

All research studies involve risks. A risk to this study you should be aware of is that some people may find the questions uncomfortable. Information obtained from this study though may help us better design interventions to address patient's unmet social needs in the future.

The results of this research study may be presented at scientific, the AMA, or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified. Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

This research study utilizes the mPATH app, a tablet-based tool, to collect study data. Dr. David Miller, a co-investigator on the study, is one of the developers of the mPATH app. Wake Forest University Health Sciences and Dr. Miller have an ownership interest in the mPATH app and could financially benefit from future sales if it is licensed for use related to this research.

| The person in charge of this study is Deepak Palakshappa. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his contact information is: |
|---|
| If you have any questions, suggestions or concerns about your rights as a volunteer in this research, contact the Institutional Review Board at 3 or the Research Subject Advocate at Wake Forest at |
| Please click the link to complete the survey. It should take less than 10 minutes to complete. By |

Please click the link to complete the survey. It should take less than 10 minutes to complete. By completing this survey, you are agreeing to participate in this study.

Thank you so much for your help,